CLINICAL TRIAL: NCT05360602
Title: Evaluation of The Effect of Alpha Lipoic Acid Administration on Oxidative Stress Markers and Occurrence of No-Reflow Phenomenon in Post Myocardial Infarction Patients
Brief Title: Alpha Lipoic Acid Effect on No-Reflow Phenomenon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omar Ragab, Dr.Omar Ragab, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NRF-123
Record Dates: First submitted 2022-04-10; First posted 2022-05-04 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: No-Reflow Phenomenon
Keywords: No-Reflow Phenomena; Alpha Lipoic Acid; Paraoxonase-1; Aldehyde dehydrogenase-2; Myocardial infarction
MeSH Terms: conditions — No-Reflow Phenomenon; Myocardial Infarction | interventions — Thioctic Acid; Dietary Supplements

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Experimental): 35 STEMI patients undergoing PCI who will receive standard of care that will include the required antiplatelet (Dual Antiplatelet Therapy; DAPT), anticoagulants, and anti-ischemic measures (high-intensity statin, ACEI, or aldosterone) as per latest guidelines recommendations.
  Interventions: Drug: The standard care for post-PCI MI
- Test group (Experimental): 35 STEMI patients undergoing PCI who will receive the standard of care in addition to IV Alpha Lipoic Acid 600 mg before PCI then 600 mg orally for 28 days after PCI
  Interventions: Dietary Supplement: Alpha Lipoic Acid plus the standard care for post-PCI MI

INTERVENTIONS:
Dietary Supplement: Alpha Lipoic Acid plus the standard care for post-PCI MI — Intravenous and oral administration of Alpha Lipoic Acid 600 mg plus the standard care for post-PCI MI which will include the required antiplatelet (Dual Antiplatelet Therapy; DAPT), anticoagulants, and anti-ischemic measures (high-intensity statin, ACEI, or aldosterone) as per latest guidelines recommendations.
  Other Names: Dietary supplement plus standard care per guidelines for post-PCI MI
  Arms: Test group
Drug: The standard care for post-PCI MI — will include the required antiplatelet (Dual Antiplatelet Therapy; DAPT), anticoagulants, and anti-ischemic measures (high-intensity statin, ACEI, or aldosterone) as per latest guidelines recommendations.
  Other Names: Guidelines MI management
  Arms: Control group

SUMMARY:
Prospective, randomized, open-label, controlled clinical trial to evaluate the efficacy and tolerability of Alpha Lipoic Acid administration on oxidative stress, inflammatory markers, clinical outcome and occurrence of No-Reflow in post myocardial infarction (MI) patients by assessment of aldehyde dehydrogenase-2 (ALDH2) as a marker of oxidative stress and paraoxonase-1 (PON-1) as a marker of oxidative stress and inflammation.

DETAILED DESCRIPTION:
All (70) STEMI patients undergoing PCI presenting to the Cardiology department will be randomly assigned into one of 2 arms: 35 patients undergoing PCI who will receive standard of care , the other 35 patients undergoing PCI will receive standard of care in addition to Alpha Lipoic Acid 600 mg daily for 4 week. IV Alpha Lipoic Acid 600 mg once daily will be administered prior to PCI then orally daily for 4 week after PCI.

Baseline evaluation included demographics and history taking. After obtaining the informed consent, information including age, weight, height, smoking state, and other diseases e.g. hypertension, diabetes, hyperlipidemias, etc. will be documented for each patient. Medication history in detail, as well as the background cardiovascular treatment, will be considered.

All patients will be followed up regularly during the hospital stay and after discharge, will be assessed for the occurrence of adverse cardiac events and occurrence of adverse effects from medications

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged >18
2. STEMI patients undergoing PCI

Exclusion Criteria:

1. Patients with a recent history of myocardial infarction (MI), a previous PCI or a previous coronary artery bypass graft
2. A late presentation (>12 h), unsuccessful primary PCI (residual stenosis >50% in the culprit lesion after procedure)
3. Pretreatment with thrombolytic or glycoprotein IIb/IIIa inhibitor therapy before primary PCI
4. Infectious or inflammatory disease
5. Severe liver or renal disease, (AST or ALT >3x ULN or Total bilirubin >2.5 x ULN), (CrCl < 60 ml/min (based on the Cockroft-Gault equation)
6. Neoplasm, or hematological disorders
7. Pregnant or breast-feeding patients
8. Active participation in another clinical study
9. Patients taking Alpha Lipoic Acid.
10. Systolic Blood pressure <90

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of No-Reflow phenomena | During 1 week post PCI
  To study the effect of Alpha Lipoic Acid administration on the occurrence of No-Reflow phenomena in post-myocardial infarction patients

SECONDARY OUTCOMES:
Evaluation of markers that reflect oxidative stress and inflammation. | Baseline, 24 hours, and 7 days post PCI
  Measuring serum concentration of aldehyde dehydrogenase-2 (ALDH2) and paraoxonase-1 (PON-1). ALDH2 reflects oxidative stress, paraoxonase-1 reflects oxidative stress and inflammation.
Occurrence of MACE. | up to 4 weeks post PCI.
  re-infarction, stroke, cardiovascular hospitalisation, and death.
Tolerability of Alpha Lipoic Acid administration | During 4 week post PCI
  Occurrence of adverse drug effects

CONTACTS AND LOCATIONS:
Overall Officials: Ayman M Saleh, MD, Study Director — Faculty of Medicine, Ain Shams University; Lamiaa M El Wakeel, PhD, Study Director — Faculty of Pharmacy, Ain Shams University; Marwa Adel Ahmed, PhD, Study Director — Faculty of Pharmacy, Ain Shams University
Locations (1):
- Ain shams hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choudhary S. Association of syntax score with short-term outcomes among acute ST-elevation myocardial infarction patients undergoing primary PCI. Indian Heart J. 2017 Apr;69 Suppl 1(Suppl 1):S20-S23. doi: 10.1016/j.ihj.2016.08.002. Epub 2016 Aug 24. PMID 28400034
- [Background] Mazhar J, Mashicharan M, Farshid A. Predictors and outcome of no-reflow post primary percutaneous coronary intervention for ST elevation myocardial infarction. Int J Cardiol Heart Vasc. 2015 Nov 6;10:8-12. doi: 10.1016/j.ijcha.2015.11.002. eCollection 2016 Mar. PMID 28616509
- [Background] Kloner RA. No-reflow phenomenon: maintaining vascular integrity. J Cardiovasc Pharmacol Ther. 2011 Sep-Dec;16(3-4):244-50. doi: 10.1177/1074248411405990. PMID 21821523
- [Background] Ndrepepa G, Tiroch K, Fusaro M, Keta D, Seyfarth M, Byrne RA, Pache J, Alger P, Mehilli J, Schomig A, Kastrati A. 5-year prognostic value of no-reflow phenomenon after percutaneous coronary intervention in patients with acute myocardial infarction. J Am Coll Cardiol. 2010 May 25;55(21):2383-9. doi: 10.1016/j.jacc.2009.12.054. PMID 20488311
- [Background] Fearon IM, Faux SP. Oxidative stress and cardiovascular disease: novel tools give (free) radical insight. J Mol Cell Cardiol. 2009 Sep;47(3):372-81. doi: 10.1016/j.yjmcc.2009.05.013. Epub 2009 May 28. PMID 19481547
- [Background] Aviram M, Rosenblat M, Bisgaier CL, Newton RS, Primo-Parmo SL, La Du BN. Paraoxonase inhibits high-density lipoprotein oxidation and preserves its functions. A possible peroxidative role for paraoxonase. J Clin Invest. 1998 Apr 15;101(8):1581-90. doi: 10.1172/JCI1649. PMID 9541487
- [Background] Wang X, Yu Y, Ji L, Liang X, Zhang T, Hai CX. Alpha-lipoic acid protects against myocardial ischemia/reperfusion injury via multiple target effects. Food Chem Toxicol. 2011 Nov;49(11):2750-7. doi: 10.1016/j.fct.2011.07.065. Epub 2011 Aug 6. PMID 21843584